CLINICAL TRIAL: NCT04536610
Title: The Effect Of Osteoporosis Education On Osteoporosis Knowledge Level and Daily Life In Parkinsonian Patients, Randomized Controlled Trial
Brief Title: Is Osteoporosis Education Effective in Parkinsonian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Selmin Gulbahar, Clinical Professor of Department of Physical Medicine and Rehabilitation, Faculty of Medicine, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Kerim OP Parkinson
Record Dates: First submitted 2020-08-25; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Osteoporosis; Parkinson Disease
Keywords: osteoporosis; parkinson disease; osteoporosis education; knowledge level; daily life
MeSH Terms: conditions — Osteoporosis; Parkinson Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Providing structured OP education in addition to the informative leaflet. (The leaflet contained the same information as the OP education program)
  Interventions: Behavioral: Providing structured osteoporosis education; Behavioral: Giving informative leaflet
- Control group (Active Comparator): Giving only the informative leaflet. (The leaflet contained the same information as the OP education program)
  Interventions: Behavioral: Giving informative leaflet

INTERVENTIONS:
Behavioral: Providing structured osteoporosis education — The OP education was performed in groups of 4-5 people by a single physician with a single session in the form of verbal expression via slide, with a duration of 20 minutes.
  Arms: Experimental group
Behavioral: Giving informative leaflet — Leaflets containe the same information as the OP education program

SUMMARY:
The effects of osteoporosis (OP) education on OP patients and the normal population studied and described in numerous studies. But the effects of OP education on Parkinsonian patients have not been sufficiently elucidated.

The purpose of this study was to evaluate the effect of OP education on the OP knowledge level and daily life in Parkinsonian patients.

Our hypothesis is; to Parkinsonian patients; there is a statistically significant difference in terms of OP knowledge level and daily life between giving only informative leaflets about OP and also providing structured OP education.

54 participants aged 50 and older with Parkinson's Disease were randomized to the experimental and control groups. While only leaflets were given to the control group, structured OP education was also given to the experimental group. Patients were evaluated with the same structured face-to-face interviews at the entrance and 12 weeks later.

DETAILED DESCRIPTION:
The OP education was performed in groups of 4-5 people by a single physician in the form of verbal expression via slide, with a duration of 20 minutes and in the form of a single session. Our leaflets contained the same information as the OP education program.

Face-to-face interviews include; Revised 2011 Osteoporosis Knowledge Test (rOKT) (0-32 points) for OP knowledge levels; National Osteoporosis Foundation daily calcium intake scale [NOF, (mg)], Physical Activity Scale For The Elderly (PASE, 0-763 points), smoking and alcohol use status (Yes/No) and quantities (cigarette pack/per week, alcohol unit/per week), frequency of falls (times/last 1 month) were questioned for effects on daily life.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 50 years or older
2. Being diagnosed with Parkinson's Disease

Exclusion Criteria:

1. Severe physical and cognitive dysability

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity Scale For The Elderly score at the endpoint | At 12th week
  (0-763 points) Higher scores mean a better outcome
National Osteoporosis Foundation daily calcium intake scale score at the endpoint | At 12th week
  (250mg - ... mg) Higher scores mean a better outcome

SECONDARY OUTCOMES:
Revised 2011 Osteoporosis Knowledge Test score at the endpoint | At 12th week
  (0-32 points) Higher scores mean a better outcome
Smoking and alcohol use status at the endpoint | At 12th week
  (Yes/No) "No" is a better status
Amount of smoking and alcohol use at the endpoint | At 12th week
  (Cigarette pack / per week, alcohol unit / per week). Lower scores mean a better outcome
Frequency of falls at the endpoint | At 12th week
  Times / last 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided